CLINICAL TRIAL: NCT05986734
Title: Evaluation of Subcutaneous Immunoglobulin Product Cutaquig in Terms of Safety and Efficacy in the Treatment of Patients With Primary Immunodeficiencies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCPHOI-2022-09
Record Dates: First submitted 2023-03-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-03

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: Primary immunodeficiency diseases; Cutaquig; intravenous immunoglobulin; subcutaneous immunoglobulin
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cutaquig — Subcutaneous immunoglobulin products are administered at the same monthly dose (0.4-0.8 g/kg), evenly divided into 3-5 administrations per month, subject to monitoring of the pre transfusion IgG level with target IgG values of at least 7 g/L.
  Other Names: subcutaneous immunoglobulin; Octapharma

SUMMARY:
In the prospective part of the study, patients diagnosed with PID will receive replacement therapy with Cutaquig for at least 6 months and will be randomised with the help of physicians of the Russian PID Registry. At the beginning of the study, data on the prior intravenous immunoglobulin (IVIG) therapy efficacy will be extracted from patients' medical records (retrospective part of study). Also, at the beginning of the study, patients or their parents will be asked to complete Quality of Life Questionnaire for children, version 4.0; short form in Russian - Pediatric Quality of Life Inventory Russian, Version 4.0 (Russia), PedSQL (Appendix 14.1). During the 6 months of treatment with Cutaquig, investigators will enter information on infectious episodes, IgG levels (at least 3 times during the study period), and definition of an adverse drug reaction / serious adverse drug reaction, in the database. After 6 months, patients/their parents will be asked to complete the PedSQL, Quality of Life Questionnaire again. If the patient continues to receive the drug, and patient and his/her legally acceptable representatives (for patients under 14 years of age) agree to continue participating in the study, similar information will be collected for another 6 months. The first 6 months are planned for the main study period, 6-12 months for an extended study period. Data obtained in the prospective phase of the study will be compared with similar data obtained in the retrospective phase in the same patients

DETAILED DESCRIPTION:
In the prospective part of the study, patients diagnosed with PID will receive replacement therapy with Cutaquig for at least 6 months and will be randomised with the help of physicians of the Russian PID Registry. At the beginning of the study, data on the prior intravenous immunoglobulin (IVIG) therapy efficacy will be extracted from patients' medical records (retrospective part of study). Also, at the beginning of the study, patients or their parents will be asked to complete Quality of Life Questionnaire for children, version 4.0; short form in Russian - Pediatric Quality of Life Inventory Russian, Version 4.0 (Russia), PedSQL (Appendix 14.1). During the 6 months of treatment with Cutaquig, investigators will enter information on infectious episodes, IgG levels (at least 3 times during the study period), and definition of an adverse drug reaction / serious adverse drug reaction, in the database. After 6 months, patients/their parents will be asked to complete the PedSQL, Quality of Life Questionnaire again. If the patient continues to receive the drug, and patient and his/her legally acceptable representatives (for patients under 14 years of age) agree to continue participating in the study, similar information will be collected for another 6 months. The first 6 months are planned for the main study period, 6-12 months for an extended study period. Data obtained in the prospective phase of the study will be compared with similar data obtained in the retrospective phase in the same patients.

Considering the lack of the study drug marketing authorisation in the Russian Federation, study drug doses and treatment regimens were chosen as per current clinical practice and instructions for human use approved in other countries. Conventionally, on switching from IVIG therapy, the subcutaneous immunoglobulin products are administered at the same monthly dose (0.4-0.8 g/kg), evenly divided into 3-5 administrations per month, subject to monitoring of the pre transfusion IgG level with target IgG values of at least 7 g/L. All this information will be reflected in the Case record forms (CRF). Besides, information about therapeutic strategies, such as dose change or therapy change, will also be entered in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over the age of 0 years with a verified diagnosis of primary immunodeficiency, who require regular immunoglobulin replacement therapy
* Patients' and/or their legal representatives' (for patients under 14 years of age) consent to participate in the study

Exclusion Criteria:

* Hypersensitivity to the study drug or any component of the study drug
* Active oncological disease
* Condition after haematopoietic stem cell transplantation
* Use of other immunoglobulin products during the study drug therapy.
* Discontinuation or irregular use of the study drug

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients diagnosed with PID. Patients of both sexes over the age of 0 years with a verified diagnosis of primary immunodeficiency, who require regular immunoglobulin replacement therapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
comparative characteristics of serum IgG concentrations in IVIG and SCIG therapy | after 3 months from the start
  analysis of the results of the study after 3 months from the start of subcutaneous immunoglobulin therapy: assessment of IgG concentration over time, box plot
Comparison of the average number of infectious complications per person per month on IVIG and SCIG therapy | after 3 months from the start
  analysis of the results of the study after 3 months from the start of subcutaneous immunoglobulin therapy: the frequency of infectious complications, box plot

SECONDARY OUTCOMES:
Pre-transfusion IgG level | 6 months from study enrollment
Frequency of unscheduled antibiotic use during the study drug therapy | 6 months from study enrollment
Duration of unscheduled antibiotic use during the study drug therapy | 6 months from study enrollment
The number of hospitalisations due to infectious diseases during the study drug therapy. | 6 months from study enrollment
Length of hospital stay due to infectious diseases during the study drug therapy | 6 months from study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Anna Shcherbina, MD,Phd, Study Director — Chief HSCT department at Federal Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No